CLINICAL TRIAL: NCT07080021
Title: A Prospective Observational Cohort Study on Longitudinal Monitoring of ctDNA MRD in Neoadjuvant Therapy for Pancreatic Cancer
Brief Title: A Cohort Study on ctDNA MRD in Neoadjuvant Therapy for Pancreatic Cancer
Acronym: MRD
Status: Recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KY01003 v2.0 /20200603
Record Dates: First submitted 2025-07-15; First posted 2025-07-23 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-05

CONDITIONS: Borderline Resectable Pancreatic Adenocarcinoma; Resectable Pancreatic Adenocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Biospecimen Retention: Samples With DNA — Specimen Type: FFPE of tumor tissue from biopsy . Whole blood samples (collected longitudinally at defined timepoints during neoadjuvant therapy and follow-up).
  Collection Purpose: NGS testing for circulating tumor DNA (ctDNA) analysis to assess Minimal Residual Disease (MRD) status.
  Collection Timeline: Before/during/after neoadjuvant therapy cycles and postoperative.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Standard Reagents, Pancreatic Cancer — This is a non-interventional study. Neoadjuvant therapy regimens and surgical approaches are determined solely by attending physicians according to clinical treatment standards.

SUMMARY:
The goal of this prospective observational study is to learn about the clinical utility of dynamic ctDNA-based Minimal Residual Disease (MRD) monitoring in patients with borderline resectable pancreatic cancer undergoing neoadjuvant therapy. The main questions it aims to answer are:

1. Does MRD negativity correlate with improved surgical outcomes (R0 resection rates) and long-term survival (Disease-Free Survival [DFS] / Overall Survival [OS])?
2. Can serial MRD status assessments guide optimal neoadjuvant therapy duration? Participants (n=119) will be adults aged 18-75 years with histologically confirmed pancreatic cancer meeting NCCN criteria for borderline resectable/high-risk resectable/locally advanced disease, deemed eligible for neoadjuvant therapy by a multidisciplinary team (MDT) and with ECOG performance status ≤1. Patients with distant metastasis, prior anticancer therapy, or concurrent malignancies are excluded.

During 24-month study period (12-month recruitment + 12-month follow-up), enrolled subjects will:

1. Receive standard-of-care neoadjuvant therapy/surgery per physician's decision.
2. Undo serial blood draws for ctDNA-MRD testing at predefined timepoints.

2. Be followed for DFS/OS outcomes for 18 months. This non-interventional study is conducted at Ruijin Hospital Pancreatic Surgery Department.

DETAILED DESCRIPTION:
Research Summary Study Name ：Prospective and Observational Study on MRD Dynamic Monitoring of Neoadjuvant Therapy for Borderline Resectable Pancreatic Cancer

Study Introduction ：This study investigates borderline resectable pancreatic cancer patients undergoing neoadjuvant therapy followed by surgical resection. It dynamically monitors Minimal Residual Disease (MRD) using circulating tumor DNA (ctDNA) technology to examine the correlation between MRD status at various monitoring points and patients' R0 resection rates, Disease-Free Survival (DFS), and Overall Survival (OS). The hypothesis states that MRD-negative patients have significantly better prognosis than MRD-positive patients.

Primary Objective ：To evaluate the correlation between ctDNA-based MRD status at different monitoring points during neoadjuvant therapy and therapeutic efficacy/prognosis (DFS/OS). To explore whether MRD status can help determine the optimal duration of neoadjuvant therapy.

Study Subjects Sample size : 119 cases

Inclusion criteria :

Age 18-75 years Pathologically confirmed pancreatic cancer Meets NCCN criteria for high-risk resectable, borderline resectable, or locally advanced disease MDT discussion confirming suitability for neoadjuvant therapy ECOG score ≤1

Exclusion criteria :

Distant metastasis History of anti-tumor therapy Concurrent other malignancies

Study Unit/Location ：Department of Pancreatic Surgery, Ruijin Hospital

Study Intervention ：This is a non-interventional study. Neoadjuvant therapy regimens and surgical approaches are determined solely by attending physicians according to clinical treatment standards.

Study Duration ：24 months (12 months recruitment + 12 months follow-up)

Subject Participation Duration ：Each subject requires 18 months to complete the study.

Protocol: A total of 119 subjects will be enrolled. Each subject will undergo 4 to 8 cycles of neoadjuvant therapy . Tumor tissue sampling will be performed once either via pre-neoadjuvant biopsy or surgical resection (biopsy-derived tissue is preferred ) and paired with serial peripheral blood sampling (for MRD detection ), as detailed in the accompanying schematic diagram.

Peripheral Blood Collection Schedule:

1. Pre-neoadjuvant treatment： End of Cycle 2 End of Cycle 3 End of Cycle 4 End of Cycle 6
2. Pre-surgery； 3.1 month Post-surgery. Sample Volume: 10 ml whole blood collected at each time point during neoadjuvant therapy; 20 ml whole blood collected at baseline (pre-treatment) , pre-surgery , and 1-month post-surgery .

Sample Handling: All collected samples will be transferred to the central laboratory for subsequent analysis. Analysis will include: high-throughput sequencing (NGS) for evaluation of Minimal Residual Disease (MRD) status .

ELIGIBILITY:
Inclusion Criteria:

* Subjects meeting ALL of the following criteria will be enrolled:

  1. Age and Gender :Aged 18-75 years, regardless of gender.
  2. Diagnosis and Disease Stage :

     Pathologically confirmed pancreatic cancer, meeting NCCN guideline criteria for:

     A. High-risk resectable (meeting ≥1 criterion):
     1. Luminal stenosis of the portal vein or superior mesenteric vein on imaging;
     2. Radiographic stage T≥3 or N≥1;
     3. Serum CA19-9 ≥1000 U/mL (after resolution of jaundice);
     4. Confirmed regional lymph node metastasis;
     5. Significant weight loss (>10% baseline) or severe pain requiring opioids.

     B. Borderline resectable :
     1. Tumor involving the common hepatic artery without celiac axis contact;
     2. Tumor contact with SMA ≤180°.

     C. Locally advanced (unresectable):
     1. Tumor encasement (>180°) of the SMA, celiac axis, or common hepatic artery;
     2. Unreconstructable involvement of SMV/portal vein;
     3. No distant metastasis.
  3. Treatment Suitability :Deemed suitable for neoadjuvant therapy after multidisciplinary team (MDT) discussion .
  4. Performance Status :ECOG (Eastern Cooperative Oncology Group) performance status ≤1 .
  5. Life Expectancy :Estimated survival ≥6 months.
  6. Organ Function :No severe cardiac, hepatic, or renal dysfunction, including:

     ALT/AST ≤3×ULN (upper limit of normal); Serum creatinine ≤1.5×ULN .
  7. Informed Consent :Signed written informed consent voluntarily provided.

Exclusion Criteria:

* Subjects meeting ANY of the following criteria will be excluded:

  1. Distant Metastasis Radiographically confirmed distant metastatic lesions.
  2. Prior Anti-Tumor Therapy History of any prior anti-tumor treatment, including:

     Systemic chemotherapy Radiotherapy Interventional therapy Immunotherapy Targeted therapy Anti-tumor traditional Chinese medicine therapy.
  3. Concurrent Malignancy Diagnosis of other active malignancies.
  4. Pregnancy or Lactation Female subjects who are pregnant or breastfeeding.
  5. Drug Allergy Hypersensitivity to any agents in the guideline-recommended first-line neoadjuvant regimen .
  6. Transplantation History Prior allogeneic hematopoietic stem cell transplantation or solid organ transplantation .
  7. Immunodeficiency Disorders Congenital or acquired immunodeficiency, including:

Human Immunodeficiency Virus (HIV) infection;

Active Hepatitis B :

HBsAg-positive andHBV-DNA ≥10,000 copies/mL (≥2,000 IU/mL) at screening;

Active Hepatitis C :

HCV-Ab-positive andHCV-RNA positive at screening; Co-infection with HBV and HC

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population consists of 119 patients aged 18-75 years with pathologically confirmed pancreatic cancer meeting NCCN-defined criteria for high-risk resectable, borderline resectable, or locally advanced stage. Eligibility requires multidisciplinary discussion (MDT) confirmation of suitability for neoadjuvant therapy, ECOG performance status ≤1, estimated survival ≥6 months, no severe organ dysfunction, and provision of informed consent. Subjects with distant metastasis, prior anti-tumor therapy, or concurrent malignancies are excluded.
Sampling Method: Non-Probability Sample
Enrollment: 119 (Estimated)
Dates: Start 2025-05-20 (Actual); Primary Completion 2026-05-20 (Estimated); Study Completion 2027-11-20 (Estimated)

PRIMARY OUTCOMES:
The correlation between ctDNA-MRD status at serial monitoring points during neoadjuvant therapy and therapeutic efficacy (R0 resection). | 1 years
  To evaluate the correlation between ctDNA-MRD status at serial monitoring points during neoadjuvant therapy and therapeutic efficacy (R0 resection).

SECONDARY OUTCOMES:
The correlation between ctDNA-MRD status at serial monitoring points during neoadjuvant therapy and survival outcomes (DFS/OS). | 2 years
  To evaluate the correlation between ctDNA-MRD status at serial monitoring points during neoadjuvant therapy and survival outcomes (DFS/OS).

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Ruijin Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai
  - Ruijin hospital, Shanghai

IPD SHARING:
Plan to Share IPD: Undecided